CLINICAL TRIAL: NCT01293006
Title: A Study to Evaluate the Effects of MK-4305 in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Suvorexant in Patients With Chronic Obstructive Pulmonary Disease (MK-4305-032)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-032
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Insomnia
Keywords: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pulmonary Disease, Chronic Obstructive | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suvorexant first, then placebo (Experimental): During Period 1, participants <65 years of age were administered a 40-mg oral dose of suvorexant once daily for 4 consecutive days in the evening and participants ≥65 years of age were administered a 30-mg oral dose of
  suvorexant once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening.
  Interventions: Drug: suvorexant; Drug: Placebo
- Placebo first, then suvorexant (Experimental): During Period 1, participants <65 years of age received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening and participants ≥65 years of age received one placebo tablet matching
  suvorexant, orally, once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants were administered a 40-mg oral dose of suvorexant once daily for 4 consecutive days in the evening.
  Interventions: Drug: suvorexant; Drug: Placebo

INTERVENTIONS:
Drug: suvorexant — one tablet (30 or 40 mg suvorexant depending on participant age: 40 mg for participants <65 years of age and 30 mg for participants ≥65 years of age), orally, once daily, for 4 consecutive days
  Other Names: MK-4305; SCH 900433
Drug: Placebo — one tablet matching suvorexant, orally, once daily, for 4 consecutive days

SUMMARY:
This study will evaluate the safety, tolerability, and effect of multiple doses of suvorexant (MK-4305) on respiratory function in participants with chronic obstructive pulmonary disease (COPD). This is a crossover study, so all participants will receive both suvorexant and placebo while on study. The primary hypothesis of this study is that multiple doses of suvorexant do not produce a clinically significant reduction of mean oxygen saturation (SaO2) during total sleep time in participants with COPD, as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential must demonstrate a serum beta-human chorionic gonadotropin (β-hCG) level consistent with the nongravid state at the prestudy (screening) visit and agree to use (and/or have their partner use) two (2) acceptable methods of birth control beginning at the prestudy visit throughout the study (including washout intervals between treatment periods/panels) and until 2 weeks after the last dose of study drug in the last treatment period. Females of non-childbearing potential (postmenopausal without menses for at least 1 year and follicle stimulating hormone [FSH] value in the postmenopausal range, or status post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy)
* Body Mass Index (BMI) ≤40 kg/m2 at the prestudy (screening)
* COPD documented by medical history and pulmonary function tests with spirometry measurements at Visit 1 meet all of the following COPD study criteria according to the modified Global Initiative for Obstructive Lung Disease (GOLD) criteria (forced expiratory volume [FEV1]/ forced vital capacity [FVC] ratio ≤70% and FEV1 ≥40% predicted [inclusive])
* Stable physical health for at least 2 weeks prior to entering the study
* No clinically significant abnormality on electrocardiogram (ECG)
* No clinically significant abnormality on the screening polysomnography (PSG) including no evidence of obstructive sleep apnea, restless leg syndrome, periodic limb movement disorder, parasomnia including nightmare disorder, sleep terror disorder and sleepwalking disorder but participants with insomnia may be enrolled
* Nonsmoker or smokes ≤20 cigarettes or equivalent per day without the urge to wake up to smoke during the night
* Sleeps for 4 hours or more per night with a usual bedtime between 8:00 post meridian (PM) and 12:30 ante meridian (AM)
* Participant must complete a sleep diary for at least 5 consecutive days and up to 21 days prior to the screening PSG visit
* Participant is reliably able to perform the study assessments; demonstrates ability to understand task instructions, and is physically capable

Exclusion Criteria:

* Participant is mentally or legally incapacitated, has significant emotional problems at the time of prestudy or expected during conduct of the study, or has a history or evidence of a clinically significant psychiatric disorder that would interfere with participation in the study
* Abnormal pre-randomization laboratory values in alanine transaminase (ALT >1.5 x the upper limit of normal [ULN]), aspartate transaminase (AST >1.5 x ULN), total bilirubin >1.5 x ULN, and serum creatinine of >2 mg/dL
* Participant has any history of a neurological disorder, including but not limited to seizure disorder (other than single episodes of childhood febrile seizures), stroke, transient ischemic attack, multiple sclerosis, cognitive impairment, or significant head trauma with sustained loss of consciousness within the last 10 years
* History of bipolar disorder, a psychotic disorder, or posttraumatic stress disorder, or psychiatric condition requiring treatment with a prohibited medication, or psychiatric condition that, in the investigator's opinion, would interfere with the patient's ability to participate in the study
* Participant has other than COPD and evidence of another clinically significant, active pulmonary disorder, such as such as bronchiectasis or asthma documented by history, physical examination, or chest x-ray
* History within the past 6 months prior to the prestudy of acute coronary syndrome, unstable angina, congestive heart failure, cardiogenic syncope, cardiomyopathy, any symptomatic arrhythmia, orthostatic hypotension, or uncontrolled hypertension
* History of neoplastic disease except adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix, malignancies which have been successfully treated ≥10 years prior to the prestudy and follow-up has revealed no evidence of recurrence from the time of treatment through the time of the prestudy, or in the opinion of the Investigator, are highly unlikely to sustain a recurrence for the duration of the study
* History or diagnosis of narcolepsy, cataplexy (familial or idiopathic), circadian rhythm sleep disorder, parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and REM behavior disorder, sleep-related Breathing Disorder (i.e., obstructive or central sleep apnea syndrome or central alveolar hypoventilation syndrome), periodic limb movement disorder, restless legs syndrome, or primary hypersomnia
* Normal PSG recording at screening
* Hematocrit > 55%
* Participant has been treated in an emergency room or has been hospitalized for COPD within 2 months prior to the screening visit, necessitating antibiotics, systemic corticosteroids, oxygen therapy
* Positive screening urine alcohol test or drug test
* Nursing mother
* Condition, therapy, lab, or ECG abnormality or other circumstances that might confound the results of the study
* Taking, or plans to take, one or more of the prohibited concomitant medications
* Participant consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages, or excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years
* Need for more than 3 toilet visits during the night
* Participant has a history of shift work (defined as permanent night shift or rotating day/night shift work) within the past 2 weeks or anticipates the need to perform shift work during the study
* Travel across 3 or more time zones (transmeridian travel) within 1 week of study start
* Participant is at imminent risk of self-harm or harm to others in the investigator's opinion
* Concerns of the investigator regarding the safe participation of the participant in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03-25 (Actual); Primary Completion 2012-01-20 (Actual); Study Completion 2012-02-22 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sun H, Palcza J, Rosenberg R, Kryger M, Siringhaus T, Rowe J, Lines C, Wagner JA, Troyer MD. Effects of suvorexant, an orexin receptor antagonist, on breathing during sleep in patients with chronic obstructive pulmonary disease. Respir Med. 2015 Mar;109(3):416-26. doi: 10.1016/j.rmed.2014.12.010. Epub 2015 Jan 5. PMID 25661282
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-032&kw=4305-032&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant (40 mg) Then Placebo: During Period 1, participants <65 years of age were administered a 40-mg oral dose of suvorexant once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening.
- Suvorexant (30 mg) Then Placebo: During Period 1, participants ≥65 years of age were administered a 30-mg oral dose of suvorexant once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening.
- Placebo Then Suvorexant (40 mg): During Period 1, participants <65 years of age received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants were administered a 40-mg oral dose of suvorexant once daily for 4 consecutive days in the evening.
- Placebo Then Suvorexant (30 mg): During Period 1, participants ≥65 years of age received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants were administered a 30-mg oral dose of suvorexant once daily for 4 consecutive days in the evening.
Period: Period 1
Arm/Group | Suvorexant (40 mg) Then Placebo | Suvorexant (30 mg) Then Placebo | Placebo Then Suvorexant (40 mg) | Placebo Then Suvorexant (30 mg)
Started | 11 | 2 | 9 | 3
Completed | 11 | 2 | 9 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Suvorexant (40 mg) Then Placebo | Suvorexant (30 mg) Then Placebo | Placebo Then Suvorexant (40 mg) | Placebo Then Suvorexant (30 mg)
Started | 11 | 2 | 9 | 3
Completed | 11 | 2 | 9 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Suvorexant (40 mg) Then Placebo | Suvorexant (30 mg) Then Placebo | Placebo Then Suvorexant (40 mg) | Placebo Then Suvorexant (30 mg)
Started | 11 | 2 | 9 | 3
Completed | 10 | 2 | 9 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Suvorexant (40 mg) Then Placebo: During Period 1, participants <65 years of age were administered a 40-mg oral dose of suvorexant once daily for 4 consecutive days in the evening. A washout period of, at least, 7 days followed Period 1. During Period 2, participants received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening.
- Suvorexant (30 mg) Then Placebo: During Period 1, participants ≥65 years of age were administered a 30-mg oral dose of MK-suvorexant once daily for 4 consecutive days in the evening. A washout period of at least 7 days followed Period 1. During Period 2, participants received one placebo tablet matching suvorexant, orally, once daily for 4 consecutive days in the evening.
- Total: Total of all reporting groups
Arm/Group | Suvorexant (40 mg) Then Placebo | Suvorexant (30 mg) Then Placebo | Placebo Then Suvorexant (40 mg) | Placebo Then Suvorexant (30 mg) | Total
Number analyzed (Participants) | 11 | 2 | 9 | 3 | 25
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [39 to 64] | 67.0 [67 to 67] | 56.7 [47 to 64] | 70.3 [69 to 72] | 58.2 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 5 | 1 | 16
  Male | 3 | 0 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Oxygen Saturation (SaO2) During Total Sleep Time
Description: Evaluation of the effect of multiple dose suvorexant (MK-4305) on SaO2 during total sleep time as measured by pulse oximetry. Lower SaO2 values are associated with sleep impairment. Total sleep time is the total of all rapid eye movement (REM) and non-REM sleep in a sleep episode.
Time Frame: Day 4 of each period
Population: Twenty-four of the 25 participants were included in the primary evaluation of SaO2 and AHI data; one participant was excluded due to a protocol violation. During the Placebo periods, there were 22 evaluable participants at Day 4; 2 participants had either no data or missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Oxygen Saturation
Groups:
- Suvorexant (30 mg or 40 mg): Participants administered either a 40-mg or a 30-mg oral dose of suvorexant.
- Placebo: Participants administered placebo.
Arm/Group | Suvorexant (30 mg or 40 mg) | Placebo
Number analyzed (Participants) | 24 | 22
Percentage of Oxygen Saturation | 93.38 [92.47 to 94.30] | 92.99 [92.06 to 93.92]
Statistical Analysis 1: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of Least Squares Means; Mean Difference (Final Values) = 0.39, 90% CI 2-sided [-0.12 to 0.91]

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 14 days after last dose
Population: All participants were included in the Safety Population.
Measure: Number; unit: participants
Groups:
- Suvorexant (40 mg): Participants administered a 40-mg oral dose of suvorexant.
- Suvorexant (30 mg): Participants administered a 30-mg oral dose of suvorexant.
Arm/Group | Suvorexant (40 mg) | Suvorexant (30 mg) | Placebo
Number analyzed (Participants) | 20 | 5 | 25
participants | 6 | 2 | 5

3. Primary Outcome: Number of Participants Discontinued From Study Drug Due to an AE
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 15 days
Population: All participants were included in the Safety Population.
Measure: Number; unit: participants
Arm/Group | Suvorexant (40 mg) | Suvorexant (30 mg) | Placebo
Number analyzed (Participants) | 20 | 5 | 25
participants | 0 | 0 | 0

4. Secondary Outcome: Percentage of Total Sleep Time in Which SaO2 is Less Than 90%, 85% or 80%
Description: Evaluation of the percentage of the night in which SaO2 is less than 90%, less than 85% and less than 80% following multiple dose administration of suvorexant and placebo. Lower SaO2 values are associated with sleep impairment.
Time Frame: Day 1 and Day 4 of each period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Total Sleep Time
Groups:
- Suvorexant (30 mg or 40 mg): Participants receiving either a 40-mg or 30-mg dose of suvorexant.
- Placebo: Participants receiving placebo.
Arm/Group | Suvorexant (30 mg or 40 mg) | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Total Sleep Time
  Day 1 (SaO2 is less than 90%) (n = 24, 24) | 6.01 [-1.48 to 13.49] | 4.98 [-2.51 to 12.46]
  Day 1 (SaO2 is less than 85%) (n = 24, 24) | 0.32 [-0.03 to 0.67] | 0.11 [-0.24 to 0.46]
  Day 1 (SaO2 is less than 80%) (n = 24, 24) | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted. | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted.
  Day 4 (SaO2 is less than 90%) (n = 24, 22) | 7.45 [0.01 to 14.89] | 6.63 [-1.05 to 14.31]
  Day 4 (SaO2 is less than 85%) (n = 24, 22) | 0.32 [0.06 to 0.58] | 0.01 [-0.26 to 0.28]
  Day 4 (SaO2 is less than 80%) (n = 24, 22) | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted. | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted.
Statistical Analysis 1: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, SaO2 <90%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Means Squares; Mean Difference (Final Values) = 1.03, 90% CI 2-sided [-1.30 to 3.36]
Statistical Analysis 2: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, SaO2 <85%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.21, 90% CI 2-sided [-0.08 to 0.50]
Statistical Analysis 3: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, SaO2 <90%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.82, 90% CI 2-sided [-5.77 to 7.41]
Statistical Analysis 4: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, SaO2 <85%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.32, 90% CI 2-sided [0.00 to 0.63]

5. Secondary Outcome: Mean Apnea/Hypopnea Index (AHI)
Description: Evaluation of the effect of multiple dose administration of suvorexant on AHI as measured by polysomnography. The AHI is an overall index of obstructive sleep apnea (OSA) severity. The AHI is calculated by dividing the number of apneas and hypopneas by the number of hours of sleep. AHI values are categorized as mild OSA = 5 to <15/hr and moderate OSA = 15 to <30/hr.
Time Frame: Day 1 and Day 4 of each period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per hour
Groups:
- Suvorexant (30 mg or 40 mg): Participants administered either a 40-mg or 30-mg dose of suvorexant.
Arm/Group | Suvorexant (30 mg or 40 mg) | Placebo
Number analyzed (Participants) | 24 | 24
Events per hour
  Day 1 (n = 24, 24) | 6.64 [4.63 to 8.66] | 5.92 [3.91 to 7.94]
  Day 4 (n = 24, 22) | 8.27 [5.71 to 10.84] | 6.22 [3.61 to 8.83]
Statistical Analysis 1: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.72, 90% CI 2-sided [-0.60 to 2.04]
Statistical Analysis 2: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 2.05, 90% CI 2-sided [0.33 to 3.77]

6. Secondary Outcome: Mean Arterial SaO2 for Different Sleep Stages
Description: Comparison of the mean SaO2 during different sleep stages (REM, Non-REM, and awake) following multiple dose administration of suvorexant and placebo. Lower SaO2 values are associated with sleep impairment. Sleep stages were determined by polysomnography.
Time Frame: Day 1 and Day 4 of each period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Oxygen Saturation
Groups:
- Suvorexant (30 mg or 40 mg): Participants administered either a 40-mg or a 30-mg dose of suvorexant.
Arm/Group | Suvorexant (30 mg or 40 mg) | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Oxygen Saturation
  Day 1 - Mean SaO2 during REM (n = 24, 24) | 93.06 [92.12 to 94.00] | 93.02 [92.08 to 93.96]
  Day 1 - Mean SaO2 during Non-REM (n = 24, 24) | 93.14 [92.26 to 94.02] | 93.27 [92.39 to 94.15]
  Day 1 - Mean SaO2 during Wake (n = 24, 24) | 94.15 [93.42 to 94.89] | 94.37 [93.63 to 95.10]
  Day 4 - Mean SaO2 during REM (n = 24, 22) | 93.21 [92.23 to 94.19] | 92.88 [91.88 to 93.87]
  Day 4 - Mean SaO2 during Non-REM (n = 24, 22) | 93.35 [92.40 to 94.30] | 93.09 [92.13 to 94.05]
  Day 4 - Mean SaO2 during Wake (n = 24, 22) | 94.31 [93.54 to 95.08] | 93.86 [93.08 to 94.64]
Statistical Analysis 1: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.41 to 0.47]
Statistical Analysis 2: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, Non-REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-0.53 to 0.27]
Statistical Analysis 3: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 1, Wake, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = -0.21, 90% CI 2-sided [-0.61 to 0.18]
Statistical Analysis 4: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [-0.32 to 0.98]
Statistical Analysis 5: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, Non-REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.26, 90% CI 2-sided [-0.26 to 0.78]
Statistical Analysis 6: Comparison: Suvorexant (30 mg or 40 mg) vs Placebo; Day 4, Wake, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [0.10 to 0.80]

7. Secondary Outcome: Mean Arterial SaO2 During Total Sleep Time
Description: Evaluation of the effect of multiple dose suvorexant on mean oxygen saturation (SaO2) during total sleep time as measured by pulse oximetry. Lower SaO2 values are associated with sleep impairment. Total sleep time is the total of all rapid eye movement (REM) and non-REM sleep in a sleep episode.
Time Frame: Day 1 of each period
Population: Twenty-four of the 25 participants were included in the primary evaluation of SaO2 and AHI data; one participant was excluded due to a protocol violation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Oxygen Saturation
Groups:
- Suvorexant (40 mg or 30 mg): Participants administered either a 40-mg or a 30-mg dose of suvorexant.
Arm/Group | Suvorexant (40 mg or 30 mg) | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Oxygen Saturation | 93.14 [92.28 to 94.00] | 93.24 [92.37 to 94.10]
Statistical Analysis 1: Comparison: Suvorexant (40 mg or 30 mg) vs Placebo; Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = -0.10, 90% CI 2-sided [-0.50 to 0.31]

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose
Groups:
- Suvorexant (40 mg): Participants administered a 40-mg dose of suvorexant.
Arm/Group | Suvorexant (40 mg) | Suvorexant (30 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/5 | 0/25
Other Adverse Events (participants affected / at risk) | 3/20 | 2/5 | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (40 mg) (N=20) | Suvorexant (30 mg) (N=5) | Placebo (N=25)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.